CLINICAL TRIAL: NCT05122156
Title: Correlation of Berg Balance Scale, Time up and Go and Dynamic Gait Index Scale in Community Dwelling Ambulatory Elderly
Brief Title: Correlation of Berg Balance Scale, Time up and Go and Dynamic Gait Index Scale in Elderly
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: RiphahIU Sajidia bibi
Record Dates: First submitted 2021-11-08; First posted 2021-11-16 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Old Age; Debility
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will find a correlation Between Berg Balance scale, Time up and Go and Dynamic Gait Index Scale in community Dwelling Ambulatory Elderly. It will be comparative cross sectional survey that will be evaluate which scale is best one for quick screening of elderly. This study will be completed within the time duration of 6 month. Convenient sampling technique will be used to collect the data. 125 sample size will be taken, in this study to find the correlation between Berg Balance scales. Time up and Go and Dynamic Gait index scale in community dwelling ambulatory elderly. In this study all subjects perform Mini-mental state examination test to meet the inclusion criteria of the study it will be above than 25 than all subjects perform Berg Balance test, Time up and Go test and Dynamic Gait Index test then interpret their values to find the best one scale for screening of elderly. . In this study subjects included will be living independently in the community and also those who walk without any aid. Those subjects who are diagnosed with neuromuscular condition, cardiorespiratory condition, cognitive impairment and having uncorrected auditory and visual deficit will be excluded from this study. In this study we will check the static, proactive part of the dynamic balance, their gait impairments and also the risk of fall of elder population. Pearson correlation Data will be analyzed on SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

65 or above 65 years old. Both male and Females. Living independently in the community. Walking without any aid. Minimental state examination score more than 25

Exclusion Criteria:

Diagnosed neuromuscular condition. Diagnosed cardiorespiratory conditions. Diagnosed cognitive impairment. Uncorrected visual and auditory deficit

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly patients more than 65 years age
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination test | Single reading
  n 1975(Folstein and McHugh) the mini-mental state test was developed and has since widely been used in clinical and research settings. This scale will be used to assess the cognition of the subjects.it is a screening tool of 30 component.
  A qualified person takes 10 minutes to complete. A score of moderate (10-20 points) and mild(21-24 points) and less than 9 score indicate significant cognitive impairment. Normal cognition is demonstrated by a score of 25 and above
Berg Balance Scale | Single reading
  Berg Balance scale is a performance-based balance test scale of 14 items. on an ordinal scale each subject is scored (0-4).Total test score range from 0(lowest ability to balance) to 56(highest balance ability.The items analyses the ability of the subject to sustain increasingly challenging positions or movements by decreasing the base of support from sitting and standing to single-leg-position
Time Up and Go test | Single reading
  Time up and go test is a successful screening method to evaluate the chance of falling. The American and British Recommendations on clinical practice Geriatric societies suggest that the TUG test be used as a primary indicator of functional assessment. Walking pace, muscle strength and balance, sit-to-walk transition time, turning, walking and walk-to-sit transition are expressed in Time Up and Go test. Participants take greater than 12 seconds to complete TUG will be at greater risk of fall
The Dynamic Gait index (DGI) | Single reading
  The Dynamic Gait index (DGI) is a method for clinical evaluation that uses a variety of gait related activities to determine the dynamic balance and risk of falling in older adults. Subjects score less than 19/24 will be at risk of falling. This scale will also be use to check the gait impairment of the elderly.

CONTACTS AND LOCATIONS:
Overall Officials: Tehreem Mukhtar, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No